CLINICAL TRIAL: NCT05526079
Title: Treatment of T2-T3/NO-N+ Adenocarcinoma of the Rectum by Neoadjuvant Chemotherapy (FOLFOX) Followed by Preoperative Chemo (Fluorouracil / Capecitabine)-Radio Therapy (CRT) With Watchful Waiting for Complete Responders
Brief Title: Watchful Waiting for Complete Responders to Therapy in Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Amr Aref, Chief of Radiation, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1291129
Record Dates: First submitted 2022-08-27; First posted 2022-09-02 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Induction FOLFOX Chemotherapy followed by concurrent chemoradiotherapy and nonoperative surveillance for complete responders
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Watchful Waiting (Experimental): Six cycles of FOLFOX (infusional fluorouracil, leucovorin, and oxaliplatin) will be administered every two weeks according to protocol. After a 3 week recovery period, this will be followed by conventional concurrent radiation and 5FU/capecitabine.
  Patients will be re-staged two to three weeks after completion of induction FOLFOX therapy to ensure no disease progression. The patients will be re-staged again at least 7-11 weeks post completion of nCRT. Patients with restaging results showing either complete or near complete response, will be allocated to "watchful waiting."
  Interventions: Other: Watchfuf waiting

INTERVENTIONS:
Other: Watchfuf waiting — Careful review of patient response with the hope of avoiding radical surgery.

SUMMARY:
The purpose of this project is to determine if in a selected group of patients, at higher risk of wound dehiscence and other complications, treatment by local excision and management by a "watchful waiting" or an initial "non-operative management" approach, with an offer of radical resection only to those patients whose tumors demonstrate "regrowth" will maintain acceptable local control and overall survival rate for the whole cohort.

DETAILED DESCRIPTION:
This is a prospective registration study of a very limited number of subjects (3-8/year) who have achieved full or near full clinical CR after neo-adjuvant FOLFOX chemotherapy prior to chemo-radiotherapy, but without subsequent surgery, to determine whether a "wait and see" approach will maintain local control while improving quality of life. Patients will undergo standard of care baseline work-up for their disease before being enrolled to the protocol followed by protocol treatment, all standard of care just in reverse order. Patients with less than 1/2 of the rectum being circumferentially involved at diagnosis will also receive additional brachytherapy which will be supported by hospital funded research dollars. Patients will undergo additional testing for study related purposes during the restaging processes such as MRI, endoscopic ultrasound, and will complete an assessment to determine impact on quality of life. Providers that will be conducting the MRI and endoscopic ultrasound have agreed to waive professional fees, as well as the hospital has agreed to waive facility fees that have been incurred while the patient is on study protocol. Patients will follow standard of care guidelines for follow up post-excision if they do not respond to treatment, and modified standard of care guidelines if their are identified as complete responders which will include additional imaging at specific milestones, again waived by providers and facility. Patients on watchful waiting, who recur locally will undergo total mesorectal excision. Patients will not be responsible for any fee incurred that is not considered standard of care.

Patients will be accrued as they present to the Van Elslander and Webber cancer center clinics. They will be enrolled in this arm of the study only if surgical evaluation indicates that surgical resection will extend to include the dentate line if said patients were candidates for local excision. We expect that about 3 patients/year will be eligible.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of rectal invasive adenocarcinoma
3. Tumor in the low rectum lying < 4 cm from the anal verge
4. Clinical stage T3/N0-N1M0.
5. Patients with low T2 who will need abdominal perineal resection are also eligible.

Exclusion Criteria:

1. Age less than 18 years
2. Other forms of cancer
3. Tumors >= 4 cm from the anal verge
4. Tumors of other clinical stages than listed above

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2028-07-09 (Estimated); Study Completion 2029-07-09 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival | three years
  Survival without recurrence of the cancer

SECONDARY OUTCOMES:
Quality of life using LARS score | three years
  Measures of patient comfort and satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Amr Aref, MD, Principal Investigator — Ascension St. John Hospital
Locations (1):
- Ascension St. John Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No